CLINICAL TRIAL: NCT01531036
Title: Imagerie 3D d'élasticité du Sein Par échographie Ultrarapide au Cours d'un Traitement Par chimiothérapie néoadjuvante.
Brief Title: 3D Breast Ultrasound Elastography in Patients Under Neoadjuvant Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: C10-02; 2010-A00663-36 (Registry Identifier: IDRCB)
Record Dates: First submitted 2012-02-08; First posted 2012-02-10 (Estimated); Last update posted 2025-08-27 (Actual); Status verified 2016-02

CONDITIONS: Malignant Breast Tumours

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- shear wave imaging (Experimental): Single arm study evaluating breast 3D elastography by means of shear wave propagation into breast tissue.
  Interventions: Device: 3D Ultrasound elastography by means of shear wave propagation into breast tissue

INTERVENTIONS:
Device: 3D Ultrasound elastography by means of shear wave propagation into breast tissue — Aixplorer Supersonic Imagine Ultrasound System with 3D probe for real-time elastography
  Other Names: Aixplorer Supersonic Imagine

SUMMARY:
Breast Ultrasound Elastography is a complementary technique permitting a better characterization of breast lesions. 3D breast ultrasound elastography is a novel technique permitting a volumetric calculation of lesion stiffness. This could be particularly useful in patients with large breast tumors under pre-operative chemotherapy

DETAILED DESCRIPTION:
3D breast ultrasound elastography provides volumetric lesion stiffness details in real time. 3D acquisition is compared to breast MRI in order to evaluate volume measurements calculated in ultrasound. Lesion elasticity is calculated in 3 planes with immediate reconstruction. The purpose of this prospective study is to evaluate the feasibility of this technique and compare the results to those of Breast MRI. For women receiving preoperative chemotherapy, this technique will be evaluated with regard to tumour shrinkage and lesion elasticity modifications under treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients having already undergone a breast MRI
* Patients presenting with breast lesions measuring between20-50mm in ultrasound

Exclusion Criteria:

* Multifocal lesions
* History of breast cancer
* Breast implants
* Inflammatory breast disease
* Pregnancy

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2010-12; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
3D volumetric elasticity measurements | 10min
  An utrafast shear wave imaging 3-plane acquisition provides several frames of breast lesion elasticity, that are reconstructed by means of a dedicated software thus permitting the direct volumetric elasticity measurements in kPa

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Athanasiou, MD, Principal Investigator — Curie Cancer Institute
Locations (1):
- Curie Cancer Institute, Paris, France

REFERENCES:
- [Background] Athanasiou A, Latorre-Ossa H, Criton A, Tardivon A, Gennisson JL, Tanter M. Feasibility of Imaging and Treatment Monitoring of Breast Lesions with Three-Dimensional Shear Wave Elastography. Ultraschall Med. 2017 Jan;38(1):51-59. doi: 10.1055/s-0034-1398980. Epub 2015 Mar 5. PMID 25741668
- [Background] Athanasiou A, Tardivon A, Tanter M, Sigal-Zafrani B, Bercoff J, Deffieux T, Gennisson JL, Fink M, Neuenschwander S. Breast lesions: quantitative elastography with supersonic shear imaging--preliminary results. Radiology. 2010 Jul;256(1):297-303. doi: 10.1148/radiol.10090385. Epub 2010 May 26. PMID 20505064